CLINICAL TRIAL: NCT05244759
Title: A Single Dose Study to Assess the Mass Balance Recovery, Absorption, Metabolism and Excretion of [14C]-BLU-5937 in Healthy Male Subjects After Oral Dosing
Brief Title: Mass Balance Recovery, Absorption, Metabolism and Excretion of [14C]-BLU-5937
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUS-P1-03
Record Dates: First submitted 2022-02-11; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Single oral dose of [14C]-BLU-5937
  Interventions: Drug: [14C]-BLU-5937

INTERVENTIONS:
Drug: [14C]-BLU-5937 — Each subject will receive a single oral administration of [14C]-BLU-5937 capsule, in the fasted state.

SUMMARY:
This is a single-centre, open-label, non-randomised, single-period, single-dose study in healthy male subjects designed to assess the mass balance recovery, PK, metabolite profile and metabolite identification of [14C]-BLU-5937.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males

Exclusion Criteria:

* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder,as judged by the investigator

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta after a single oral dose of [14C]-BLU-5937 | 168 hour
  Mass balance recovery of total radioactivity in all excreta by analysing the total radioactivity and metabolic profile in blood, urine and faeces samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: No